CLINICAL TRIAL: NCT02013050
Title: A Phase 2,Double-Blind, Randomized, Placebo-Controlled, Dose Escalating, Multicenter Study of SGX942 For the Attenuation of Oral Mucositis in Patients Being Treated With Concomitant Chemoradiation for the Treatment of Squamous Cell Carcinoma of the Head and Neck
Brief Title: A Dose Escalating Study of SGX942 for Oral Mucositis in Patients With Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Soligenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDR-OM-01
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Control
  Interventions: Drug: Placebo
- SGX942 (Experimental): Investigational Drug i) 1.5 mg/kg ii) 3.0 mg/kg iii) 6.0 mg/kg
  Interventions: Drug: SGX942

INTERVENTIONS:
Drug: SGX942
  Arms: SGX942
Drug: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of SGX942 in patients receiving chemoradiation treatment for the treatment of head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven non-metastatic squamous cell carcinoma of the mouth or oropharynx and is planned to receive a standard course of concomitant CRT.
* Patients who have received surgery are eligible if surgery is performed within 6 weeks prior to study initiation.
* Planned to receive standard cisplatin chemotherapy administered either weekly or every third week.
* Must be able to read and understand informed consent
* Adequate birth control methods for the duration of the study

Exclusion Criteria:

* Current mucositis.
* Prior radiation to the head and neck.
* Chemotherapy treatment within the previous 12 months.
* Tumors of the lips, sinuses, salivary glands or nasopharynx.
* Unknown primary tumor.
* Stage 4c metastases.
* Evidence of significant hepatic, hematologic, or immunologic disease.
* Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Markey Cancer Center-University of Kentucky, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients were randomized but never received study drug and are excluded from the analyses
Groups:
- Placebo; 1.5 mg/kg; 3.0 mg/kg; 6.0 mg/kg: Administered as a 4-minute intravenous (IV) infusion, every 3 days (±1 day) while receiving radiation therapy to a maximum of 14 doses
Period: Overall Study
Arm/Group | Placebo | 1.5 mg/kg | 3.0 mg/kg | 6.0 mg/kg
Started | 42 | 41 | 3 | 23
Completed | 38 | 36 | 3 | 19
Not Completed | 4 | 5 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 1.5 mg/kg | 3.0 mg/kg | 6.0 mg/kg | Total
Number analyzed (Participants) | 42 | 41 | 3 | 23 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 2 | 20 | 84
  >=65 years | 11 | 10 | 1 | 3 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 2 | 3 | 23
  Male | 33 | 32 | 1 | 20 | 86
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 3 | 6
  Not Hispanic or Latino | 40 | 38 | 3 | 20 | 101
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 2 | 5 | 0 | 2 | 9
  White | 38 | 36 | 3 | 20 | 97
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 41 | 3 | 23 | 109

OUTCOME MEASURES:

1. Primary Outcome: Duration of Severe Oral Mucositis (SOM)
Description: Duration of SOM was defined as the number of days from the onset of SOM until resolution of SOM. If the patient did not meet the requirements for resolution of SOM by the 1-month follow up visit, he/she was considered censored at the 1-month follow-up visit (or point of discontinuation of the study, if the patient had discontinued prior to the end of planned treatment). Patients who did not experience SOM were assigned a duration of 0.01. OM was evaluated using the published World Health Organization (WHO) OM grading scale that uses a scale of 0 to 4.
Time Frame: 4 weeks after end of therapy
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | 1.5 mg/kg | 3.0 mg/kg | 6.0 mg/kg
Number analyzed (Participants) | 38 | 36 | 3 | 19
days | 18 [5 to 36] | 9 [3 to 19] | 14 [0 to NA] — The sample size does not allow | 22 [3 to 36]

2. Secondary Outcome: Residual Severe Oral Mucositis (SOM)
Description: OM was evaluated using the published World Health Organization (WHO) OM grading scale that uses a scale of 0 to 4. SOM is defined as a WHO score of greater than or equal to 3.
Time Frame: 4 weeks after end of therapy
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1.5 mg/kg | 3.0 mg/kg | 6.0 mg/kg
Number analyzed (Participants) | 38 | 36 | 3 | 19
percentage of participants | 21 | 6 | 33 | 16

3. Secondary Outcome: Duration of Severe Oral Mucositis (SOM)
Description: as for outcome 2
Time Frame: 4 weeks after end of therapy
Measure: Median (95% Confidence Interval); unit: WHO score * days
Arm/Group | Placebo | 1.5 mg/kg | 3.0 mg/kg | 6.0 mg/kg
Number analyzed (Participants) | 38 | 36 | 3 | 19
WHO score * days | 35.5 [0 to 222] | 21.8 [0 to 210] | 33.0 [0 to 84] | 46.5 [0 to 167]

4. Secondary Outcome: Incidence of Clinically Reported, Non-fungal Infections
Time Frame: 4 weeks after end of therapy
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1.5 mg/kg | 3.0 mg/kg | 6.0 mg/kg
Number analyzed (Participants) | 38 | 36 | 3 | 19
percentage of participants | 45 | 28 | 0 | 21

5. Secondary Outcome: Percent of Patients With RECIST 1.1 Classification of "Complete Response"
Description: The RECIST 1.1 scoring system evaluates both the defined (target) tumor, the non-target lesions, and the appearance of new lesions on radiologic scans as follows:
  Target Lesion :
  Complete Response (CR): All target lesions gone Partial Response (PR): >30% decrease from Baseline Progressive Disease (PD): >20% increase from smallest sum of longest diameter recorded since treatment started (best response) Stable Disease (SD): Neither PD nor PR
  Non-Target Lesion:
  Complete Response (CR): All non-target lesions gone,Tumor markers gone Stable Disease (SD): Persistence of ≥1 non-target lesion, Tumor marker level elevated Progressive Disease: Enlargement of non-target lesions
Time Frame: 4 weeks after end of therapy
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1.5 mg/kg | 3.0 mg/kg | 6.0 mg/kg
Number analyzed (Participants) | 38 | 36 | 3 | 19
percentage of participants | 39 | 47 | 33 | 21

6. Secondary Outcome: Duration of Severe Oral Mucositis (SOM) in Patients Receiving Every 3rd Week Cisplatin
Time Frame: 4 weeks after end of therapy
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | 1.5 mg/kg | 3.0 mg/kg | 6.0 mg/kg
Number analyzed (Participants) | 22 | 24 | 3 | 10
days | 30 [5 to 65] | 10 [0 to 19] | 14 [0 to NA] — The sample size does not allow | 17 [0 to NA] — The sample size does not allow

7. Secondary Outcome: Incidence of Severe Oral Mucositis (SOM) in Patients Receiving Every 3rd Week Cisplatin
Time Frame: 4 weeks after end of therapy
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1.5 mg/kg | 3.0 mg/kg | 6.0 mg/kg
Number analyzed (Participants) | 22 | 24 | 3 | 10
percentage of participants | 82 | 67 | 67 | 80

8. Secondary Outcome: Survival
Time Frame: 12 months after end of therapy
Population: Safety Population: all patients randomized who received at least 1 dose of study drug and were included in the dose group of the drug that they actually received instead of the drug dose they were randomized. 2 patients were randomized but never received drug and are excluded. 1 patient was randomized to placebo but received 1.5 mg/kg SGX942.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1.5 mg/kg | 3.0 mg/kg | 6.0 mg/kg
Number analyzed (Participants) | 43 | 41 | 3 | 24
percentage of participants | 81 | 93 | 100 | 83

9. Secondary Outcome: Percent of Patients With RECIST 1.1 Classification of "Complete Response"
Description: as for outcome 5
Time Frame: 12 months after end of therapy
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 1.5 mg/kg | 3.0 mg/kg | 6.0 mg/kg
Number analyzed (Participants) | 38 | 36 | 3 | 19
percentage of participants | 53 | 53 | 33 | 53

ADVERSE EVENTS:
Time Frame: From the time of enrollment up until four weeks (±5 days) following the last study drug treatment.
Description: Safety analyses were performed on the Safety Population which is comprised of all patients randomized who received at least 1 dose of study drug and were included in the dose group of the drug they actually received instead of the drug dose to which they were randomized. 2 patients were randomized but never received drug and are excluded from the analyses. 1 patient was randomized to placebo but received 1.5 mg/kg SGX942 and is included in the 1.5 mg/kg treatment group in all safety analyses.
Arm/Group | Placebo | 1.5 mg/kg | 3.0 mg/kg | 6.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 8/43 | 3/41 | 0/3 | 4/24
Serious Adverse Events (participants affected / at risk) | 25/41 | 25/42 | 1/3 | 16/23
Other Adverse Events (participants affected / at risk) | 41/41 | 42/42 | 3/3 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | 1.5 mg/kg (N=42) | 3.0 mg/kg (N=3) | 6.0 mg/kg (N=23)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3
White blood cell disorder (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 2 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Feeding tube complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 4 | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal disorder (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Peripheral artery thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | 1.5 mg/kg (N=42) | 3.0 mg/kg (N=3) | 6.0 mg/kg (N=23)
Anaemia (Blood and lymphatic system disorders) | 5 | 13 | 1 | 6
Blood disorder (Blood and lymphatic system disorders) | 2 | 2 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 3
Neutrophil function disorder (Blood and lymphatic system disorders) | 2 | 4 | 1 | 3
Platelet disorder (Blood and lymphatic system disorders) | 5 | 7 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 3
White blood cell disorder (Blood and lymphatic system disorders) | 6 | 16 | 1 | 6
Atrial fibrillation (Cardiac disorders) | 0 | 3 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 2 | 1 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 1
Tinnitus (Ear and labyrinth disorders) | 9 | 6 | 0 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 23 | 18 | 2 | 11
Diarrhea (Gastrointestinal disorders) | 6 | 10 | 0 | 3
Dry mouth (Gastrointestinal disorders) | 11 | 14 | 2 | 7
Dyspepsia (Gastrointestinal disorders) | 7 | 4 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 11 | 14 | 3 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3 | 0 | 3
Gingival pain (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 29 | 31 | 3 | 20
Odynophagia (Gastrointestinal disorders) | 4 | 6 | 0 | 3
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 3 | 2 | 0 | 4
Oral pain (Gastrointestinal disorders) | 10 | 5 | 0 | 2
Saliva altered (Gastrointestinal disorders) | 2 | 3 | 1 | 1
Salivary duct inflammation (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Vomiting (Gastrointestinal disorders) | 15 | 23 | 2 | 12
Asthenia (General disorders) | 2 | 3 | 0 | 1
Chills (General disorders) | 2 | 2 | 2 | 2
Fatigue (General disorders) | 21 | 23 | 2 | 12
Malaise (General disorders) | 0 | 1 | 0 | 2
Medical device complication (General disorders) | 3 | 0 | 0 | 0
Oedema peripheral (General disorders) | 5 | 3 | 0 | 1
Pyrexia (General disorders) | 6 | 12 | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 4 | 1 | 0
Candida infection (Infections and infestations) | 7 | 8 | 0 | 3
Fungal infection (Infections and infestations) | 3 | 1 | 0 | 1
Oral candidiasis (Infections and infestations) | 6 | 12 | 1 | 1
Pneumonia (Infections and infestations) | 3 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 0 | 2
Radiation skin injury (Injury, poisoning and procedural complications) | 10 | 14 | 1 | 6
Abnormal loss of weight (Metabolism and nutrition disorders) | 8 | 13 | 2 | 10
Decreased appetite (Metabolism and nutrition disorders) | 12 | 10 | 1 | 9
Dehydration (Metabolism and nutrition disorders) | 10 | 17 | 0 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 5 | 0 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 3 | 4 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 7 | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 7 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 11 | 1 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 10 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 9 | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3
Ageusia (Nervous system disorders) | 3 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 6 | 8 | 1 | 3
Dysgeusia (Nervous system disorders) | 11 | 22 | 2 | 13
Headache (Nervous system disorders) | 6 | 12 | 1 | 2
Syncope (Nervous system disorders) | 0 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 4 | 2 | 0 | 4
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 2
Depression (Psychiatric disorders) | 1 | 1 | 0 | 4
Insomnia (Psychiatric disorders) | 6 | 4 | 1 | 5
Proteinuria (Renal and urinary disorders) | 1 | 3 | 1 | 0
Renal disorder (Renal and urinary disorders) | 4 | 7 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 3 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0 | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 17 | 2 | 8
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 5 | 6 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 | 5 | 0 | 1
Hypertension (Vascular disorders) | 3 | 7 | 1 | 2
Hypotension (Vascular disorders) | 2 | 6 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There were limitations put on the sites from publishing data until the sponsor had published data. That data is now published.